CLINICAL TRIAL: NCT04953507
Title: Evaluation of T2, T3 Sympathectomy for Postmastectomy Pain Syndrome by Thermal Radiofrequency Versus Chemical Neurolysis Using Perfusion Index Derived Pulse Oximeter
Brief Title: Evaluation of T2, T3 Sympathectomy for Postmastectomy Pain Syndrome by Pulse Oximeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2104-50104
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Transurethral Resection of Prostate; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Radiofrequency (Experimental): T2, T3 block by thermal radiofrequency lesioning at 80°c for 120 seconds
  Interventions: Procedure: Thermal Radiofrequency
- Chemical Neurolysis (Active Comparator): T2, T3 block by chemical neurolysis using 1.5 ml of phenol in saline 8% at each level
  Interventions: Procedure: Chemical Neurolysis

INTERVENTIONS:
Procedure: Thermal Radiofrequency — Radiofrequency lesioning at level of T2 and T3 using 80°c for 120 seconds
  Arms: Thermal Radiofrequency
Procedure: Chemical Neurolysis — injection of 1.5 ml of the chemical neurolytic agent (phenol in saline 8%) at each level
  Arms: Chemical Neurolysis

SUMMARY:
The aim of the study is to compare the efficacy of T2, T3 sympathetic block using thermal radiofrequency versus chemical neurolysis in postmastectomy pain syndrome using perfusion index derived from pulse oximetry.

DETAILED DESCRIPTION:
Postmastectomy pain is a chronic pain condition with neuropathic nature. Several drugs and methods are used for its management. This study was designed to compare the efficacy of both thermal radiofrequency and chemical neurolysis in management of postmastectomy pain through using perfusion index derived from pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with postmastectomy pain syndrome
* ≥ Age 18 years
* ASA II-III

Exclusion Criteria:

* patient refusal
* coagulation defects
* abnormal kidney or liver functions
* local infection at site of injection
* bone metastases
* severe cardiorespiratory disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | up to 24 weeks
  minimum score 0 and maximum score 10

SECONDARY OUTCOMES:
Perfusion index trend | procedure time
  measuring the change in perfusion index in the ipsilateral limb after the procedure compared to pre-procedural
Opioid consumption | up to 24 weeks
  average opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant Professor of Anesthesia and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be available upon reasonable request through contacting the corresponding author